CLINICAL TRIAL: NCT05396547
Title: Study On The Performance And Safety Of The REVISYON SDS 100 Device On Visual Acuity In Subjects With Cataract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edinburgh Biosciences Ltd (Industry)
Collaborators: MDX Research (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EB-CE-01
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Age-related Cataract
Keywords: non-invasive cataract treatment, N-LOCS III grade 1 to 3
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Single arm interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated (Experimental): Treatment with REVISYON SDS 100 Device
  Interventions: Device: Treated with REVISYON SDS 100 Device

INTERVENTIONS:
Device: Treated with REVISYON SDS 100 Device — Treated with REVISYON SDS 100 Device

SUMMARY:
Single arm, unmasked study to evaluate the performance and safety of the REVISYON SDS 100 Device for the non-invasive treatment of vision loss in age-related cataract.

DETAILED DESCRIPTION:
This single arm, unmasked study will evaluate the performance and safety of the REVISYON SDS 100 Device for the non-invasive treatment of vision loss in age-related cataract.

Only one of the subject's eyes will be treated with the REVISYON SDS 100 Device during the study (blue light treatment beam: Visit 1: 15 minutes, Visits 2 - 9: 20 minutes). The Treatment period will last 19 days (+ 1 day), starting with the day of first treatment (Visit 1, day 1). During this period, subjects will be treated with the REVISYON SDS 100 investigational device three-times a week for 3 weeks (Visit 1 to Visit 9) up to a maximum of 20 days (or 2.9 weeks). The Treatment period will be followed by 84 days (± 10 days) of follow up, up to a maximum of 94 days (or 13.4 weeks).

The subject's eyes will be examined throughout the study to allow safety and performance to be monitored. The safety examinations includes standard ophthalmological tests.

Clinical assessments in the study will use traditional ophthalmic methods including LogMAR best corrected visual acuity (BCVA) for distance, and grading of cataracts using LOCS III.

In addition, spectral data (fluorescent emission) will be collected using the REVISYON SDS 100 Device to monitor the progress of the treatment, and to determine the suitability of these measurements for future clinical diagnoses.

ELIGIBILITY:
Inclusion Criteria:

1. Subject diagnosed with nuclear sclerotic (NS) lens opacities cataract, LOCS III grade 1 to 3 (moderate), as confirmed by the Investigator
2. Subject aged between 40 and 85 years of age (inclusive) at the time of consent
3. Best Corrected Visual Acuity (BCVA) of 0.3 LogMAR or worse due to cataract only
4. Subject whom the medical health history has been reviewed by the Investigator and medical records do not contraindicate the participation to the study
5. Subject who is judged suitable for the study after ophthalmic examination carried out by the Investigator
6. Be able and willing to follow instructions, including participation in all study assessments and visits, according to the opinion of the investigator - including being able to sit upright for at least 20 mins (duration of the treatment)

Exclusion Criteria:

1. Subject unable to give voluntary written informed consent, is unlikely to cooperate or is legally incompetent, including subjects who are institutionalised by court or official order, or in a dependency relationship with sponsor, testing centre or investigator
2. Subject who had been clinically diagnosed with any eye diseases which may impact upon the treatment, or the subject's ability to be assessed after treatment
3. Subjects with intraocular lens (IOL) implant in either eye
4. Planned replacement of crystalline lens with intraocular lens (IOL) implant within the planned study period
5. Subject with shallow anterior chamber
6. Subject who have had a fluorescence angiogram or any use of fluorescein within the last 3 days
7. Subject presenting eye infection or eye damage in either eye
8. Any condition which could interfere with the subject's ability to comply with the study including participation in all study assessments and visits.
9. Subject who had undergone a treatment using photodynamic drugs within the last 30 days. (Including but not limited to methylene blue, toluidine blue, Visudyne®, Foscan, Photofrin or 5-aminolevulinic acid/ALA)
10. Subject diagnosed with any other health condition which, in the opinion of the Investigator, would pose a safety risk to the subject by participating in the study, or may interfere with or jeopardise the study evaluation, procedures or completion
11. Subject currently receiving treatment in another investigational study or has completed another investigational study within the last 30 days
12. Subject participated in the previous study with the REVISYON Device (EB-14-LAT)
13. Females who are pregnant or lactating
14. Females who are of childbearing potential (menses within the last 12 months) and not taking adequate contraceptive precautions are excluded from the trial. Females of childbearing potential taking acceptable contraceptive precautions may be included.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Change in Visual Acuity | 4 weeks
  Change in Best Corrected Visual Acuity (BCVA), assessed using LogMAR scale.

SECONDARY OUTCOMES:
Change in Cataract Severity | 4 weeks
  Change in Cataract Severity, assessed using LOCS III
Subjective satisfaction using Visual Function Index | 4 weeks
  Subjective satisfaction, assessed using Visual Function Index (VF-14). The total result per subject is divided by the maximum possible result, excluding questions marked as "N/A," to determine the differences between the VF-14 result at Visit 1 and the VF-14 result at Visit 10. Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Shields, Study Director — Edinburgh Biosciences Ltd
Locations (11):
- Latvia (3):
  - Lens-L Ltd, Liepāja
  - Dr.Solomatina Acu Centrs, Riga
  - Zielmelkurzeme Regional Hospital, Ventspils
- Lithuania (2):
  - The Hospital of Lithuanian University of Health Sciences (LSMU) Kauno klinikos, Department of Ophthalmology, Kaunas
  - Vilnius University Hospital Santaros Klinikos, Center of Eye Diseases, Vilnius
- Romania (6):
  - Spitalul Clinic de Urgențe Oftalmologice, Depatement of Ophthamology, Bucharest
  - Vedis Ophthalmology Clinic | Ophthalmological Center Dr. Samoila, Cluj-Napoca
  - Opticlass Ophthalmology Clinic, Timișoara
  - CF Timisoara Clinical Hospital, Timișoara
  - Clinica de Oftalmologie Dr. Berghian, Timișoara
  - Clinica Vista, Ophtalmology Department, Timișoara

IPD SHARING:
Plan to Share IPD: No